CLINICAL TRIAL: NCT01690637
Title: Efficacy of Early Oseltamivir Phosphate Treatment at Hospital Admission to Reduce Severity of Illness Among Children Aged Less Than 10 Years Hospitalized With Influenza in El Salvador and Panama
Brief Title: Panama and El Salvador Children's Oseltamivir Study
Acronym: PECOS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slower than anticipated participant accrual
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Universidad del Valle, Guatemala (Other); Hospital Nacional San Juan de Dios de Santa Ana, El Salvador (Unknown); Hospital Nacional San Juan de Dios de San Miguel, El Salvador (Unknown); Hospital Del Nino, Panama (Unknown); Hospital de Especialidades Pediátricas Omar Torrijos Herrera, Panama (Unknown); Hospital Jose Domingo de Obaldia, Panama (Unknown)
Responsible Party: Principal Investigator, Fatimah Dawood, Medical Epidemiologist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDC-NCIRD-6330
Record Dates: First submitted 2012-09-17; First posted 2012-09-24 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Influenza; Human Influenza
Keywords: Oseltamivir; Tamiflu
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oseltamivir phosphate suspension (Active Comparator): Participants assigned to the oseltamivir phosphate treatment arm will receive the appropriate weight-based dose of oseltamivir phosphate every 12 hours for 10 doses. For children 0-11 months of age, oseltamivir phosphate will be dosed as 3mg/kg/dose every 12 hours. For children 12 months and older, oseltamivir phosphate will be dosed as follows: 30 mg every 12 hours for children up to 15kg, 45mg every 12 hours for children greater than 15kg up to 23 kg, 60mg every 12 hours for children greater than 23 up to 40kg, and 75mg every 12 hours for children greater than 40kg.
  Interventions: Drug: Oseltamivir phosphate suspension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir phosphate suspension
  Other Names: Tamiflu
  Arms: Oseltamivir phosphate suspension
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled trial that will be conducted in tertiary care pediatric hospitals in El Salvador and Panama. The primary purpose of this study is to determine whether empiric oseltamivir phosphate treatment given at the time of hospital admission to children less than 10 years of age hospitalized with influenza can effectively reduce their illness severity. Additional objectives are to: 1) evaluate the tolerability of oseltamivir phosphate treatment, 2) evaluate the effect of oseltamivir treatment on viral clearance and development of oseltamivir-resistant influenza virus during and after treatment in children hospitalized with influenza, 3) estimate the direct and indirect costs of all-cause respiratory illness and influenza-associated respiratory illness requiring hospitalization, and 4) evaluate the effect of empiric oseltamivir treatment during the influenza season on these costs.

The primary study hypothesis is that children with laboratory-confirmed influenza receiving empiric oseltamivir phosphate treatment initiated at the time of hospital admission will have a shorter duration of hospitalization and a shorter time to resolution of signs of severe respiratory illness compared to children receiving placebo. The secondary study hypotheses are that children with laboratory-confirmed influenza receiving oseltamivir phosphate treatment will have a reduction in the time to non-detectable influenza virus and influenza viral RNA and children with all-cause respiratory illness receiving oseltamivir phosphate will not be more likely to experience severe adverse events than children receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age <10 years
* Accompanied by a parent or guardian who has the capacity to grant and sign the written informed consent and who has consented to enrollment
* Has respiratory illness as defined by modified IMCI criteria for pneumonia:
* Cough or sore throat AND Fast breathing, defined as respiratory rate 60 breaths per minutes or greater for children 0 to <2 months, OR respiratory rate 50 breaths per minute or greater for children 2 to <12 months, OR respiratory rate 40 breaths per minute or greater for children 12 to <60 months, OR respiratory rate 30 breaths per minute or greater for children 5-9 years
* Planned for hospital admission

Exclusion Criteria:

* Symptom onset 7 days or more at the time of study screening where day 1 is the day of symptom onset
* Concomitant severe vomiting illness prior to enrollment that would preclude ability to take medication orally defined as more than 3 vomiting episodes in the preceding 24 hours
* Prematurity (birth at less than 37 weeks gestation) for children aged less than 3 months
* Birth weight less than 2500 grams for children aged less than 3 months
* Chronic supplemental oxygen requirement at home
* Known history of renal dysfunction
* History of gastrointestinal resection resulting in gastrointestinal abnormality that might hinder absorption of oral medication (such as short-gut syndrome)
* History of previous serious adverse reaction to oseltamivir phosphate
* Receipt of oseltamivir phosphate during the 5 days prior to presentation at the admitting hospital
* Previous enrollment in this study during a hospitalization that ended less than 14 days prior to the current admission

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 721 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | Participants will be followed for the duration of hospital stay, an expected median of 7 days
  Day 1 is defined as the day of arrival at the emergency department
Time to resolution of increased work of breathing | Participants will be followed for the duration of hospital stay, an expected median of 7 days
  Increased work of breathing is defined as presence of 1 or more of the following: supraclavicular retractions, subcostal or intercostal retractions, nasal flaring, grunting, or need for noninvasive or invasive mechanical ventilation, and resolution is defined as 12 hours or more without increased work of breathing in a child with increased work of breathing at enrollment
Time to resolution of hypoxia | Participants will be followed for the duration of hospital stay, an expected median of 7 days
  Hypoxia is defined as O2 saturation less than 92% measured by pulse oximetry while breathing room air or need for noninvasive or invasive mechanical ventilation and resolution is defined as 12 hours or more without hypoxia in a child with hypoxia at enrollment

SECONDARY OUTCOMES:
Incidence of new onset respiratory failure 24 hours or more after first dose of study medication | Participants will be followed for the duration of hospital stay, an expected median of 7 days
  Respiratory failure is defined by need for noninvasive or invasive mechanical ventilation
Incidence of admission to intensive care unit 24 hours or more after first dose of study medication | Participants will be followed for the duration of hospital stay, an expected median of 7 days
Incidence of death 24 hours or more after first dose of study medication | Participants will be followed up through 7 days after hospital discharge
Time to non-detectable influenza virus by viral culture and non-detectable influenza viral RNA by RT-PCR | Participants will be followed for the duration of hospital stay (an expected median of 7 days) or up through 21 days of hospitalization, whichever is shorter
Proportion of children with oseltamivir resistant virus detected during or after oseltamivir phosphate treatment who had oseltamivir susceptible virus infection at enrollment | Participants will be followed for the duration of hospital stay (an expected median of 7 days) or up through 21 days of hospitalization, whichever is shorter
Proportion of participants experiencing adverse events (including severe and non-severe) | Up through 7 days after hospital discharge
  An adverse event is defined as any unfavorable or undesirable effect (sign, symptom, abnormality, or condition), regardless of causal relationship to study procedures or participation that occurs in participants while enrolled in this clinical trial. Any medical condition or sign/symptom that is present at the time the participant is screened is considered as baseline and not reported as an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah S Dawood, MD, Principal Investigator — Centers for Disease Control and Prevention; Jorge Jara, MD, Principal Investigator — Universidad del Valle, Guatemala
Locations (5):
- El Salvador (2):
  - Hospital Nacional San Juan de Dios de San Miguel, San Miguel
  - Hospital Nacional San Juan de Dios de Santa Ana, Santa Ana
- Panama (3):
  - Hospital Jose Domingo de Obaldia, David
  - Hospital de Especialidades Pediátricas Omar Torrijos Herrera, Panama City
  - Hospital Del Nino, Panama City

REFERENCES:
- [Derived] Jara JH, Azziz-Baumgartner E, De Leon T, Luciani K, Brizuela YS, Estripeaut D, Castillo JM, Barahona A, Corro M, Cazares R, Vergara O, Rauda R, Gonzalez R, Franco D, Widdowson MA, Clara W, Alvis-Estrada JP, Murray CT, Ortega-Sanchez IR, Dawood FS. Costs associated with acute respiratory illness and select virus infections in hospitalized children, El Salvador and Panama, 2012-2013. J Infect. 2019 Aug;79(2):108-114. doi: 10.1016/j.jinf.2019.05.021. Epub 2019 May 31. PMID 31153920